CLINICAL TRIAL: NCT02271854
Title: A Randomized, Double-blind, Placebo-controlled, Within-subject Study to Evaluate the Efficacy and Safety of Diclofenac Sodium Topical Gel (DSG) 1% Applied Four Times Daily in Subjects Experiencing Acute Delayed Onset Muscle Soreness (DOMS) of the Lower Limbs
Brief Title: A Within-subject Study to Evaluate the Efficacy and Safety of Diclofenac Sodium Topical Gel 1% Compared to Placebo in Subjects Experiencing Delayed Onset Muscle Soreness
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 197-P-323
Record Dates: First submitted 2014-10-20; First posted 2014-10-22 (Estimated); Results first posted 2016-04-05 (Estimated); Last update posted 2016-04-05 (Estimated); Status verified 2016-03

CONDITIONS: Muscle Soreness
MeSH Terms: conditions — Myalgia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- diclofenac sodium gel 1% (Experimental): diclofenac sodium gel 1% applied four times daily
  Interventions: Drug: Diclofenac sodium gel 1%; Drug: Placebo
- Placebo (Placebo Comparator): Placebo gel applied four times daily
  Interventions: Drug: Diclofenac sodium gel 1%; Drug: Placebo

INTERVENTIONS:
Drug: Diclofenac sodium gel 1% — Diclofenac sodium gel 1% four times daily (This study is a within-subject design i.e. active drug applied to one leg and placebo to the other leg at the same time. Therefore the study design is not a cross-over).
Drug: Placebo — Placebo gel four times daily (This study is a within-subject design i.e. active drug applied to one leg and placebo to the other leg at the same time. Therefore the study design is not a cross-over).

SUMMARY:
This study will assess the analgesic efficacy of DSG 1% compared to placebo in the reduction of the pain associated with DOMS

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged 18-35 years
* Not engaged in regular lower extremity fitness activities in the past 6 months prior to screening
* Willing to refrain from use of ice, heat and massage during the study
* DOMS score ≥4 Pain at Rest (PAR) and a DOMS score ≥5 Pain on Walking (POW), with moderate or severe on categorical scale

Exclusion Criteria:

* Pain medication & corticosteroids prior to randomization
* Topical analgesic or anti-inflammatory treatment over the previous month
* Body mass index of >32 kg/m2

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2014-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Lotus Clinical Research, 100 W California Blvd,, Pasadena, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study Start 7 Oct 2014 and End 24 dec 2014
Groups:
- Diclofenac Sodium Gel 1% and Placebo Gel: This study is a within-subject design i.e. diclofenac sodium gel 1% four times a day applied to one leg and placebo gel four times a day applied to the other leg to the other leg at the same time
Period: Overall Study
Arm/Group | Diclofenac Sodium Gel 1% and Placebo Gel
Started | 102
Completed | 98
Not Completed | 4
Not completed — Withdrawal by Subject | 2
Not completed — Unable or unwilling to cooperate with st | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: ITT population: All randomized subjects who received at least one dose of the study drug on both legs = 102 Modified ITT population: Excludes the first 16 subjects who were systematically underdosed =86 Safety population: All randomized subjects who received at least one dose of study drug on either leg =102
Groups:
- Diclofenac Sodium Gel 1%: diclofenac sodium gel 1% applied four times daily
  Diclofenac sodium gel 1%: Diclofenac sodium gel 1% four times daily
Arm/Group | Diclofenac Sodium Gel 1%
Number analyzed (Participants) | 86
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.5 (4.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37
  Male | 49
Region of Enrollment [Number; unit: participants]
  United States | 86

OUTCOME MEASURES:

1. Primary Outcome: Sum of Pain Intensity Differences Over 24 Hours After Initiating Treatment (SPID 24), Derived From POW.
Description: The primary efficacy outcome was the time-weighted SPID 24 (POW). Sum of pain intensity differences over 24 hours after initiating treatment (SPID 24) for the modified ITT population. SPID 24 derived from Pain on Walking (POW) scores assessed over 24 hours on a 0 (No pain) - 10 (Pain as bad as you can imagine) Numerical Rating Scale. SPID 24 was computed using the trapezoidal rule, i.e. Σ [T(i) - T(i-1)] x [((PID)(i-1) + PID(i))/2] in an obvious notation, where T(i) is nominal time and PID(i), the pain intensity difference at Time i, is the baseline pain intensity (PI) score - PI score at Time i.
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: units on a scale (NRS)
Groups:
- Placebo: Placebo gel applied four times daily
  Diclofenac sodium gel 1%: Diclofenac sodium gel 1% four times daily
Arm/Group | Diclofenac Sodium Gel 1% | Placebo
Number analyzed (Participants) | 86 | 86
units on a scale (NRS) | 50.15 (35.95) | 54.83 (37.04)

2. Secondary Outcome: Sum of Pain Intensity Differences Over 48 Hours After Initiating Treatment (SPID 48), Derived From POW.
Description: Sum of pain intensity differences over 48 hours after initiating treatment (SPID 48) (POW) was a secondary outcome.
  Sum of pain intensity differences over 48 hours after initiating treatment (SPID 48) for the modified ITT population. SPID 48 derived from Pain on Walking (POW) scores assessed over 48 hours on a 0 (No pain) - 10 (Pain as bad as you can imagine) Numerical Rating Scale. SPID 48 was computed using the trapezoidal rule, i.e. Σ [T(i) - T(i-1)] x [((PID)(i-1) + PID(i))/2] in an obvious notation, where T(i) is nominal time and PID(i), the pain intensity difference at Time i, is the baseline pain intensity (PI) score - PI score at Time i.
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: units on a scale (NRS)
Arm/Group | Diclofenac Sodium Gel 1% | Placebo
Number analyzed (Participants) | 86 | 86
units on a scale (NRS) | 151.8 (81.9) | 160.84 (83.15)

ADVERSE EVENTS:
Arm/Group | Diclofenac Sodium Gel 1%
Serious Adverse Events (participants affected / at risk) | 0/102
Other Adverse Events (participants affected / at risk) | 0/102

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Preliminary agreement between Novartis Consumer Health and the investigator